CLINICAL TRIAL: NCT06323889
Title: Longitudinal Monitoring During Different Intermittent Fasting Protocols in Obese Adults - a Randomized Clinical Trial
Brief Title: Longitudinal Monitoring During Intermittent Fasting Protocols in Obese Adults
Acronym: LIMITFOOD2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIMITFOOD2
Record Dates: First submitted 2024-03-06; First posted 2024-03-21 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Intermittent Fasting; Obesity; Time Restricted Eating
Keywords: Overnutrition; Nutrition Disorders; Body Weight; Obesity; Longitudinal monitoring
MeSH Terms: conditions — Intermittent Fasting; Obesity; Overnutrition; Nutrition Disorders; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Modified Alternate Day Fasting (mADF) (Active Comparator): Participants in the mADF group will be instructed to eat every second-day ad libitum ("feast days"), and to consume a very low carbohydrate snack, restricted to the evening, provided by the study team and to otherwise abstain from calorie intake on the rest of the fast day.
  Interventions: Behavioral: Modified Alternate Day Fasting
- Time-Restricted Eating (TRE) (Active Comparator): TRE participants are instructed to eat two main meals and limit snacking from 12:00 to 20:00 daily, and to fast from 20:00 until 12:00 daily
  Interventions: Behavioral: Time-Restricted Eating
- Control group (Other): The control group will receive guidance on a quantitative reduction in total caloric intake by following a balanced diet, but no timing window for food intake will be prescribed to the participants in the control group.
  Interventions: Behavioral: Weight-loss counseling

INTERVENTIONS:
Behavioral: Modified Alternate Day Fasting — Participants are instructed to fast every other day.
  Arms: Modified Alternate Day Fasting (mADF)
Behavioral: Time-Restricted Eating — Participants are instructed to limit food intake to two main meals consumed in maximum 8 hours per day
  Arms: Time-Restricted Eating (TRE)
Behavioral: Weight-loss counseling — Participants will receive nutrition counseling to structure their main meals according to the plate model for weight-loss and to reduce number of consumed plates.
  Arms: Control group

SUMMARY:
LIMITFOOD2 is a randomized clinical intervention study that investigates the effects of two different intermittent fasting protocols compared to a control group on the health of obese adults. A total of 90 participants will be randomized into three equally sized groups: a modified alternate day fasting, a time-restricted eating and a control group, receiving general weight-loss counseling.

DETAILED DESCRIPTION:
The prevalence of overweight and obesity worldwide has risen considerably in the past century with more than one billion overweight persons, and about 600 million obese patients in 2015. Humans in modern societies typically eat at least three main meals per day and snacks around the clock. This change in eating pattern in terms of quantity and frequency leads to overconsumption of food and consequently to excess weight. Furthermore, obesity increases the risk of developing diabetes, cardiovascular disease and several types of cancer. The world health organization (WHO) has stated that there are 2.8 million deaths per year as a result of overweight and obesity.

In recent years, the concept of re-introduced fasting intervals in the form of intermittent fasting (IF) protocols became a popular alternative dietary strategy with the aim to achieve weight control and improve metabolic health. There are several different IF protocols, the most popular is time-restricted eating (TRE), which allows ad libitum (at one's pleasure) energy intake within a defined time period each time (6 to 12 hours). Another IF protocol is alternate day fasting (ADF), on 'feast days' one can consume food ad libitum, while on 'fast days' no or little food is consumed, feast and fast days alternate throughout the week. Animal studies and previous human clinical trials have provided evidence that various types of IF lead to weight loss and improved health markers. So far, interventional studies focused on the comparison of IF versus a control group, however only few studies compared different IF protocols directly. Given both the evidence for beneficial effects of IF as well as its growing popularity, it seems mandatory to reveal possible differences in the effectiveness of different protocols.

The present project will allow to directly compare two types of IF with each other and with a control group in obese participants. Furthermore, established and novel monitoring tools to track individual progress during IF are scarcely used so far but may become an important help in the future and thus, will be implemented in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-50 years, both inclusive
* Obese, BMI between 30 and 40 kg/m^2 (obesity grade I or II), both inclusive
* Non-smoker
* Good knowledge of German or English language
* Stable weight change (change < +/- 3% current bodyweight) for 3 months prior to the study
* HbA1c < 6.5% without glucose lowering medication
* LDL-cholesterol < 4.6mmol/l without lipid lowering medication

Exclusion Criteria:

* Participants who have a fasting period of > 12h per day on a regular basis and do not eat at least three main meals per day.
* Current habitual use of dietary supplements (e.g., vitamins, minerals) and/or unwillingness to cease intake of dietary supplements.
* Antibiotics intake during 3 months prior to the study due to possible interference with metabolic parameters
* Food intolerances, allergies and sensitivities (severe food allergies) or dietary restrictions (e.g. vegan lifestyle)
* Acute or chronic infections, malignant disease, renal, hepatic (more than two-fold increased transaminases), pulmonary, neurological (epilepsy) or psychiatric diseases, manifested atherosclerosis, or any other disease precluding participation in the study.
* Diabetes
* Known alcohol, substance or drug abuse, concomitant medication
* More than four hours of physical exercise per week
* Women who are pregnant, breast-feeding or aiming to become pregnant during course of the trial
* Women and men on hormonal supplementation
* Women with an irregular menstrual cycle according to the FIGO criteria
* Therapy with antidepressants within the past 6 months
* Regular therapy with acetylsalicyclic acid or current medication to regulate blood sugar, blood pressure or lipids
* Participants likely to fail to comply with the study protocol
* Participants who do not give informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Fat Volume | 8 weeks
  Change in body fat volume measured with MRI

SECONDARY OUTCOMES:
Distribution of fat volume | 8 weeks
  Changes in subcutaneous and visceral fat volume measured with MRI
Concentration of Leptin | 8 weeks
  Change in leptin concentrations will be measured.
Changes in Insulin Sensitivity | 8 weeks
  Insulin Sensitivity will be assessed using the homeostasis model assessment of insulin resistance (HOMA-IR), which is calculated from insulin and glucose concentration from a 12 hours fasting blood sample.
Changes in Fasting Lipids | 8 weeks
  Changes in concentration of Apolipoprotein B and triglycerides will be measured from a 12 hours fasting blood sample.
Changes in Inflammatory Markers | 8 weeks
  Changes in concentration of C-reactive protein and Interleukin-1beta will be measured.
Free triiodothyronine (fT3) | 8 weeks
  Change in serum levels of fT3 will be measured.

OTHER OUTCOMES:
Correlation of longitudinally measured parameters | 8 weeks
  Breath acetone measurements and continuous glucose monitoring will be conducted and correlated to the fat volume change.
Serum Metabolomics | 8 weeks
  Metabolomics provides an insight into the organisms current metabolite profile. Exploring the effect of intermittent fasting on specific metabolites could provide important insights.
Genetic Analysis | 8 weeks
  Genes associated with obesity could have an effect on the efficacy of the intermittent fasting intervention and genetic analysis may provide an important step towards personalized medicine.
LDL Particle Size | 8 weeks
  Changes in serum LDL particle size might be measured.
Fecal Microbiome | 8 weeks
  Sequencing will be used to identify the composition of bacteria and archaea within the fecal samples. Exploring the changes in the microbiome induced by intermittent fasting could provide valuable insights.

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Gerber, MD, Principal Investigator — University of Zurich
Locations (1):
- Department of Endocrinology, Diabetology and Clinical Nutrition, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No